CLINICAL TRIAL: NCT04743219
Title: Selective Removal Technique With or Without the Use of a Bioactive Material for the Management of Deep Caries Lesions in Permanent Posterior Teeth With Close Apex. A Randomized Clinical Trial.
Brief Title: Selective Removal Technique With or Without a Bioactive Material for Deep Caries Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Patricia Terceño Jiménez, DDS, MS, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0212202023220
Record Dates: First submitted 2021-02-01; First posted 2021-02-08 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Deep Caries
MeSH Terms: interventions — tricalcium silicate

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodentine Group (Active Comparator): Biodentine group: patients with mature permanent posterior teeth with deep caries lesions treated with the selective removal technique to soft dentin with Biodentine as indirect pulp capping material before placement of a definitive direct composite resin restoration.
  Interventions: Procedure: Selective removal to soft dentin, Biodentine
- No base Group (Experimental): The experimental group or No Base group: patients with mature permanent posterior teeth with deep caries lesions treated with the selective removal technique to soft dentin without the placement of a bioactive material as a base and restored directly with a definitive direct composite resin restoration.
  Interventions: Procedure: Selective removal to soft dentin, No Base

INTERVENTIONS:
Procedure: Selective removal to soft dentin, Biodentine — Carious tissue removed until its complete elimination from the lateral walls of the cavity using a round tungsten carbide bur at low speed until consistency of hard dentin around perimeter. With a manual excavator, the central cariogenic biomass will be removed, specifically the superficial part of the necrotic and demineralized caries dentin.
  In the Biodentine group, Biodentine (Septodont) will be placed on the base of the cavity with a thickness of 2 mm.
  The last step will be to perform a definitive direct resin restoration according to clinical indication.
  Arms: Biodentine Group
Procedure: Selective removal to soft dentin, No Base — Carious tissue removed until its complete elimination from the lateral walls of the cavity using a round tungsten carbide bur at low speed until consistency of hard dentin around perimeter. With a manual excavator, the central cariogenic biomass will be removed, specifically the superficial part of the necrotic and demineralized caries dentin.
  In the No base group, no bioactive material will be placed as a liner, the 3M Scothcbonf Universal Plus adhesive will be placed directly over the remaining dentin surface.
  The last step will be to perform a definitive direct resin restoration according to clinical indication.
  Arms: No base Group

SUMMARY:
Objectives: To evaluate and compare clinical and radiographic success of the selective removal to soft dentine technique in one step using calcium silicate cement (Biodentine) vs. no indirect pulp capping material in patients with deep caries lesions in mature permanent posterior teeth with normal or reversible pulpitis after a 2 year follow-up. Evaluate the integrity of the resin composite restorations using FDI criteria.

Material and methods: selective removal to soft dentine in one visit will be performed in 104 blinded patients that will be randomly allocated into 2 study arms, 52 patients will constitute the Biodentine group and 52 the No material group. Clinical examination will be performed to obtain pre-, intra- and postoperative data, including vitality test results, periapical status and risk of caries of the patients. Periapical and bitewing radiographs will be taken before treatment (T-0), at 1 month (T-1), 6 months (T-2), 12 months (T-3) and 24 months (T-4). Restorations will be assessed using the FDI criteria at the same follow up periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 15 years.
* Parents or guardians of patients under 18 years of age, but over 15 years of age, and patients over 18 years of age who demonstrate understanding of the study and willingness to participate as evidenced by signing the voluntary informed consent and who receive a signed and dated copy of the informed consent form.
* Occlusal or occlusal-proximal caries lesions, Class I or Class II, in molars or premolars with enamel margins and affecting maximum one proximal wall.
* Molar or premolar with deep caries lesion, involving equal to or greater than two thirds of dentin in depth, with a radiographically identifiable band of healthy dentin separating the pulp chamber roof from the caries lesion.
* Normal response to tests of sensitivity (normal pulp) or discomfort when cold stimulus is applied that disappears in a couple of seconds after the elimination of the stimulus (reversible pulpitits).
* Teeth with negative percussion.

Exclusion Criteria:

* Patients immunosuppressed or with severe systemic diseases.
* Teeth with root or cervical resorption.
* Teeth with obliteration of the pulp chamber.
* Periapical or furcal radiolucency.
* Patients with periodontal disease.
* Patients with spontaneous acute pain, prolonged excruciating pain and / or pain that disturbs night sleep.
* Patients who have an allergy to any of the materials used in the treatment.
* Patients with caries lesions that during the treatment of their removal a pulp exposure is performed.
* Patients with inadequate initial radiographs for analysis.
* Evidence of pre-cancerous or cancerous lesions.
* Patients who have taken antibiotics in the last two weeks.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 2 years
  Clinical success is defined as healthy pulp, determined by a normal positive not prolonged response in the clinical examination to the cold test and the electrical test, negative response to percussion, absence of symptoms or signs of infection (abscess, fistula, swelling or inflammation) and absence of spontaneous pain.

SECONDARY OUTCOMES:
Radiographic success | 2 years
  Radiographic success is defined as the absence of widening of the periodontal ligament space (twice the equivalent of the adjacent healthy tooth) and the absence of a periapical or furcal lesion on radiographic examination. A periapical lesion is considered to be a radiolucency associated with the radiographic apex of the root of a size greater than twice the width of the periodontal ligament space.

OTHER OUTCOMES:
Failure composite resin restorations | 2 years
  FDI criteria will be used to assess the integrity of the composite resin restorations,It will be considered a restoration failure when the restoration presents a property classified as clinically unsatisfactory or poor. Thus, body fracture or loss of restoration, damage to the margin, weak contact point or food impaction, marginal or large gap, secondary caries or if the patient is not satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ceballos, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No